CLINICAL TRIAL: NCT04732585
Title: Kinematic Assessment of Real-Time Motion Acquisition of the Human Lower Limb Peripheral Joints by Dynamic 4D Transversal Imaging (KARMA-4D)
Brief Title: Kinematic Assessment of Human Peripheral Joints by Dynamic CT
Acronym: Karma-4D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Johan de Mey, Prof. dr. Johan de Mey, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.U.N 143201733617
Record Dates: First submitted 2021-01-21; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Patellofemoral Pain Syndrome; ACL Tear
Keywords: Dynamic CT; Kinematics; Patellofemoral pain syndrome; Rehabilitation; Surgery; ACL reconstruction
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Anterior Cruciate Ligament Injuries | interventions — Physical Therapy Modalities; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Study on PFPS patients:
  Non-randomized Controlled clinical trial
  Study on ACL patients:
  Non-randomized Controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with PFPS or ACL injury (Experimental): Physiotherapy intervention Surgical intervention
  Interventions: Procedure: Physiotherapy or Surgery
- Healthy control group (No Intervention): The healthy control group will not do any intervention

INTERVENTIONS:
Procedure: Physiotherapy or Surgery — Physiotherapy: Guidelines suggest a tailored and progressive exercise program to improve muscle strength and control, joint mobility, and patient understanding of the problem and how to manage it. Additional interventions like tape or manual treatment can also be implemented but should not be exclusive
  Surgery: ACL surgical reconstruction
  Arms: Patient with PFPS or ACL injury

SUMMARY:
Aim of the research project:

The entire research project aims to investigate human peripheral joints (knee, foot & ankle, elbow, wrist & hand) by dynamic 4D radiographic imaging acquisition during real-time motion.

Aim of the specific study on Patellofemoral pain syndrome (PFPS) patients:

This study aims to investigate kinematics and motion changes pre and post physiotherapy intervention in patients with patellofemoral pain syndrome (PFPS) and compare them with a healthy control group.

Aim of the specific study on patients undergoing ACL reconstruction:

This study aims to investigate kinematics and motion changes pre and post-surgical intervention in patients with ACL injury that require surgical reconstruction and compare them with a healthy control group.

DETAILED DESCRIPTION:
Study on PFPS patients:

Non-randomized Control Clinical Trial. The patient that satisfies inclusion and exclusion criteria is informed about the nature study at the orthopaedic outpatient clinic. If necessary, the study coordinator provides additional information to the patient. Informed consent will be obtained prior to inclusion in the study. The patient will be asked to undergo a dynamic scan of the knees prior to and after the physiotherapy treatment. The physiotherapy treatment is not specifically controlled but best evidence-based guidelines are provided to the patient's physiotherapist in order to have an intervention as homogeneous as possible. Guidelines suggest a tailored and progressive exercise program to improve muscle strength and control, joint mobility, and patient understanding of the problem and how to manage it. Additional interventions like tape or manual treatment can also be implemented but should not be exclusive. During imaging acquisition, the patients lay on the CT's bed with the lower limb inside the gantry. They are asked to perform a repetitive movement of the knee into different planes of motion (i.e. flexion-extension). Before the start of the dynamic CT scan protocol, a physical examination is performed by a physiotherapist. It consists of muscle strength (dynamometer) and joint ROM assessment. VAS scale and Kujala and KOOS questionnaires will be also administrated to the patients. Healthy volunteers will be provided with a brief explanation of the study the moment they make contact to be involved. Further information and informed consent will be obtained on the day of the scan. Identical procedure for the CT scan and physical assessment used with the patient will be used for the healthy subjects.

Study on patients with ACL injury:

Non-randomized Control Clinical Trial. The patient that satisfies inclusion and exclusion criteria is informed about the nature study at the orthopaedic outpatient clinic. If necessary, the study coordinator provides additional information to the patient. Informed consent will be obtained prior to inclusion in the study. The patient will be asked to undergo a dynamic scan of the knees prior to and approximately 6 weeks after ACL surgical reconstruction. Type of surgical intervention is on surgeon discretion following Best-Evidence practice guidelines.

During imaging acquisition, the patients lay on the CT's bed with the lower limb inside the gantry. They are asked to perform a repetitive movement of the knee into different planes of motion (i.e. flexion-extension). Before the start of the dynamic CT scan protocol, a physical examination is performed by a physiotherapist. It consists of muscle strength (dynamometer) and joint ROM assessment. VAS scale and Lysholm and IKDC questionnaires will be also administrated to the patients. Healthy volunteers will be provided with a brief explanation of the study the moment they make contact to be involved. Further information and informed consent will be obtained on the day of the scan. Identical procedure for the CT scan and physical assessment used with the patient will be used for the healthy subjects.

ELIGIBILITY:
Study patient with PFPS:

Inclusion Criteria:

patellar/anterior knee pain, provoked by functional activities such as Squatting, Ascending/Descending stairs, Prolonged sitting, Kneeling, Jumping and/or running.

Exclusion Criteria:

* Metallic implants in the proximity of the knee.
* Affections of the Central Nervous System, including Cerebellar dysfunction, Stroke, ALS and MS, affect the strength, motor control and/or coordination of human joints and produce "abnormal" movement patterns;
* Affections of the Peripheral Nervous System of the lower limb, including Lumbar radiculopathy, Peripheral nerve entrapment and Neuropathy, affect the proprioception and muscle force.
* Pregnant women.
* Inflammatory Conditions
* Hyperlaxity
* Patella Dislocation
* knee injection less than 3 months

Study patient with ACL injury:

Inclusion Criteria:

ACL that requires surgical reconstruction. Imaging findings of ACL injury (MRI)

Exclusion Criteria:

* Metallic implants in the proximity of the knee.
* Affections of the Central Nervous System, including Cerebellar dysfunction, Stroke, ALS and MS, affect the strength, motor control and/or coordination of human joints and produce "abnormal" movement patterns;
* Affections of the Peripheral Nervous System of the lower limb, including Lumbar radiculopathy, Peripheral nerve entrapment and Neuropathy, affect the proprioception and muscle force.
* Pregnant women.
* Inflammatory Conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change of the amount of Rotation of knee joint (degrees) | Change from Baseline at 1-3 weeks after the end of physiotherapy intervention
  Rotations calculated as Cardan angles, rotation around the axis of rotation, Lateral Tilt of the Patella
Change of the amount of Rotation of knee joint (degrees) | Change from Baseline at 6 weeks after surgical intervention
  Rotations calculated as Cardan angles, rotation around the axis of rotation, Lateral Tilt of the Patella
Change of the amount of Translation of knee joint (mm) | Change from Baseline at 1-3 weeks after the end of physiotherapy intervention
  Translation of individual bones, translation of the axis of rotation and tibial-tuberosity to trochlear groove distance
Change of the amount of Translation of knee joint (mm) | Change from Baseline at 6 weeks after surgical intervention
  Translation of individual bones, translation of the axis of rotation and tibial-tuberosity to trochlear groove distance

SECONDARY OUTCOMES:
Change of Pain assessed by Numeric Pain Rating scale (NPRS) | Change from Baseline at 1-3 weeks after the end of physiotherapy intervention
  Patient choose between 0-10 integers that best reflects the intensity of the pain
Change of Pain assessed by Numeric Pain Rating scale (NPRS) | Change from Baseline at 6 weeks after surgical intervention
  Patient choose between 0-10 integers that best reflects the intensity of the pain
Change of Pain assessed by Numeric Pain Rating scale (NPRS) | Change from Baseline at 6 and 12 months post surgical or physiotherapy intervention
  Patient choose between 0-10 integers that best reflects the intensity of the pain
Change of Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from Baseline at 1-3 weeks after the end of physiotherapy intervention
  It is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
Change of Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from Baseline at 6 and 12 months post physiotherapy intervention
  It is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
Change of Kujala or Anterior Knee Pain Scale (AKPS) | Change from Baseline at 1-3 weeks after the end of physiotherapy intervention
  13 questions on the Kujala questionnaire total to 100 points.
Change of Kujala or Anterior Knee Pain Scale (AKPS) | Change from Baseline at 6 and 12 months post physiotherapy intervention
  13 questions on the Kujala questionnaire total to 100 points.
Change of Lysholm score | Change from Baseline at 6 weeks after surgical intervention
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting
Change of Lysholm score | Change from Baseline at 6 and 12 months post surgical intervention
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting
Change of International Knee Documentation Committee Subjective Knee Form (IKDC) | Change from Baseline at 6 weeks after surgical intervention
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items)
Change of International Knee Documentation Committee Subjective Knee Form (IKDC) | Change from Baseline at 6 and 12 months post surgical intervention
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items)

CONTACTS AND LOCATIONS:
Overall Officials: Johan de Mey, Prof, Principal Investigator — universitair ZB
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No